CLINICAL TRIAL: NCT05632666
Title: Respiratory Muscle Training in Patients With Spinal Muscular Atrophy (SMA).
Acronym: RESISTANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Princess Beatrix Muscle Foundation (Other)
Responsible Party: Principal Investigator, Dr. H.J. (Erik) Hulzebos, Clinical exercise physiologist, Child Development and Exercise Center, Wilhelmina Children's Hospital, University Medical Center Utrecht, PO Box 85090, 3508 AB, Utrecht, The Netherlands, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: W.OB19-01
Record Dates: First submitted 2022-11-02; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; Inspiratory Muscle Training; Expiratory Muscle Training; Maximum Inspiratory Mouth Pressure; Maximum Expiratory Mouth Pressure; Respiratory Muscle Training
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Inhalation

STUDY DESIGN:
Intervention Model Description: In the first four months of the study, the active treatment group will receive inspiratory muscle training starting at a therapeutic intensity of 30% of maximum inspiratory mouth pressure (PImax) and expiratory muscle training starting at a therapeutic intensity of 30% of maximum expiratory mouth pressure (PEmax). The sham-control group will receive the same training protocol but with a low (10% of PImax and PEmax) non-therapeutic intensity.
  After four months, the sham-control group will also be provided with a supervised RMT at a therapeutic intensity of 30% of PImax and PEmax.
Who Masked: Outcomes Assessor
Masking Description: The lung function analyst is blinded for treatment allocation. A data analyst will design and sign the data analysis plan in advance. The data will be analyzed according to the analysis plan by a physiotherapist who is not blinded for treatment allocation. The physiotherapists who will perform the two-weekly telephone calls are not blinded for treatment allocation. Patients will know that there are two treatment groups, and they are informed that it is not yet known which treatment is most effective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment group (Experimental)
  Interventions: Other: Inspiratory and expiratory muscle training at a therapeutic intensity
- Sham-controlled group (Sham Comparator)
  Interventions: Other: Inspiratory and expiratory muscle training at a non-therapeutic intensity

INTERVENTIONS:
Other: Inspiratory and expiratory muscle training at a therapeutic intensity — The active treatment group will receive inspiratory muscle training starting at a therapeutic intensity of 30% of maximum inspiratory mouth pressure (PImax) and expiratory muscle training starting at a therapeutic intensity of 30% of maximum expiratory mouth pressure (PEmax) for 4 months.
  In the active treatment group, the inspiratory and expiratory threshold (intensity) will be adjusted to the perceived exertion (measured with a Borg scale).
  Arms: Active treatment group
Other: Inspiratory and expiratory muscle training at a non-therapeutic intensity — The sham-control group will receive the same training protocol as the active treatment group but with a low (10% of PImax and PEmax) and stable non-therapeutic intensity.
  Arms: Sham-controlled group

SUMMARY:
The goal of this clinical trial is to study respiratory muscle training in patients with Spinal Muscular Atrophy (SMA). The main questions it aims to answer are:

* Is a home-based individualized training program for the inspiratory and expiratory muscles feasible (good adherence and good acceptability)?
* Can a home-based individualized training program for the inspiratory and expiratory muscles increase the strength of these muscles? Participants will be asked to perform 10 training sessions per week, spread out over 5-7 days. Each training session consists of 30 breathing cycles through the inspiratory muscle trainer and 30 breathing cycles trough the expiratory muscle trainer.

In the first four months of the study researchers will compare two groups to see if a higher trainings load is more effective.

One group will start at a trainings load of 10% of their maximal inspiratory and expiratory muscle strength.

The other group will start at a trainings load of 30% of their maximal inspiratory and expiratory muscle strength. This group also need to adjust the trainings load based on their perceived exertion.

After four months all participants will train on a trainings load of 30% of their maximal inspiratory and expiratory muscle strength and adjust the trainings load based on their perceived exertion.

The participants will come to the hospital for lung function tests every four months for 12 months.

DETAILED DESCRIPTION:
The aim of this study is to assess the feasibility and efficacy of respiratory muscle training in patients with SMA and respiratory muscle weakness. The hypothesis is that an individualized incremental home-based respiratory muscle training program will be feasible and will improve inspiratory muscle strength, expiratory muscle strength, lung function and patient reported breathing difficulties in patients with SMA.

Study setting: This study is conducted at the outpatient department of the Netherlands SMA center and the Child Development and Exercise Center at the University Medical Center Utrecht (UMCU), The Netherlands. All members of the study team, consisting of physicians, physiotherapists, lung function technicians, clinical exercise physiologists and nurses, have broad experience with SMA due to the national cohort study that is carried out in this center since 2010.

Study design: The RESISTANT study is an investigator-initiated, mono-center study consisting of two parts:

Part 1 (0-4 months): a single blinded randomized sham-controlled trial (RCT). In the first part of the study, the feasibility and efficacy of respiratory muscle training (RMT) in patients with SMA will be determined.

Before the first visit, participants will be recruited for enrollment by a research nurse. Patients who express interest in participating receive a patient information letter and an appointment with the physiotherapist. At the first visit (M0), the physiotherapist further determines whether patients are eligible for participation. After signing the informed consent form, participants are weighed and their length is determined, followed by lung function tests. If the maximum inspiratory mouth pressure (PImax) >80 centimeter of Water Column (cmH2O), participants are excluded for the study. If PImax ≤ 80 cmH2O, participants will be stratified prior to randomization based on PImax (group 1: PImax <60 cmH2O, group 2: PImax ≥60 cmH2O, 60 cmH2O was the median PImax in the group of patients used for the natural history study). Participants will be randomly allocated to the intervention or sham-control group. A variable block randomization method with allocation concealment in a centralized system will be used for randomization. The lung function analyst is blinded for treatment allocation. A data analyst will design and sign the data analysis plan in advance. The data will be analyzed according to the analysis plan by a physiotherapist who is not blinded for treatment allocation. The physiotherapists who will perform the two-weekly telephone calls are not blinded for treatment allocation. Patients will know that there are two treatment groups, and they are informed that it is not yet known which treatment is most effective.

All participants (and parents) will be instructed by a trained physiotherapist on the use of both devices at the first visit (baseline or M0). Participants are instructed to aim for 10 training sessions per week, divided over 5 to 7 days. A minimum of 6 hours in between training sessions is recommended. Per training session, the participant breathes 30 times through the POWERbreathe (inspiratory muscle training) and 30 times through the reverse Threshold® IMT (expiratory muscle training). If necessary, the participant may take a break, with a maximum of 60 seconds after 10 or 15 breaths. After each session they fill in a diary, which contains information about the load and the perceived exertion (Borg scale 0-10).

In the active treatment group, the intensity of the training is set at M0 at 30% of PImax and maximum expiratory mouth pressure (PEmax) and will be increased or decreased based on level of perceived exertion. Participants are instructed to increase the intensity with 1-5 cmH2O if they score a perceived exertion of 0-4 and decrease the intensity if they score a perceived exertion of 7-10. If they score a perceived exertion of 5 or 6, the intensity will not me adjusted. The intensity of the training in the sham-controlled group will be set at M0 at 10% of PImax and PEmax and will remain the same during the first 4 months of training.

- Inspiratory muscle trainer: For the inspiratory muscle training (IMT) the Conformité Européenne certified POWERbreathe KHP2 is used. Clinical research has shown high participant motivation and adherence to training with the POWERbreathe KHP2 thanks to the on-screen feedback. Furthermore, healthcare professionals can review participant progress by tracking up to 30 of the participants training sessions which the KHP2 is able to store. This data can be scrolled through to monitor progress. The electronic, variable, tapered flow valve ensures maximum training benefit. It is easy to use, easy to clean and training improvements can be easily monitored.

- Expiratory muscle trainer: For the expiratory muscle training (EMT) the Threshold Inspiratory Muscle Trainer (IMT) (Philips Respironics) in reverse is used. Use of the Threshold Positive Expiratory Pressure (PEP) (Philips Respironics) is one method to perform EMT. However, the maximal expiratory resistance of the Threshold PEP is limited to 20 cmH20. To overcome this limitation in expiratory resistance, the Threshold IMT will be used in reverse. This device contains, at its end, a valve closed by the positive pressure of a spring, which can be graded from 9 to 41 cmH2O and allows resistance changes by 1 cmH2O increments. The reverse Threshold IMT has a one-way spring-loaded valve, that closes during expiration and requires that participants exhale hard enough, to open the valve and let the air go out. This device provides constant pressure for expiratory muscle training, regardless of how quickly or slowly the participant breathes, and the optimal loading pressure can be adjusted, based upon the individual characteristics of the participant.

Part 2 (5-12 months): open label extension phase. In the second part of the study, the sham-control group will be provided with a supervised RMT at a therapeutic intensity of 30% of PImax and PEmax and the long-term effects of RMT on the occurrence of respiratory infections, health related quality of life and feasibility will be investigated in the active treatment and sham-controlled group.

Participants will visit our outpatient department every 4 months for 12 months after inclusion for assessment of primary and secondary outcome measures. This study is currently ongoing; the first participant was included on 2-2-2021. Study completion is expected in the first quarter of 2023.

Sample size: Based on a previous report on inspiratory muscle training in patients with neuromuscular diseases (n=27, 18 patients with Duchenne Muscular Dystrophy (DMD) and 9 patients with SMA) indicating a mean improvement in PImax of 28 cmH2O difference (SD ±26.27), a mean difference of 20 cmH2O (SD 25.0) is assumed between active and sham treated patients after 4 months. To detect this effect size with 80% power and two-sided alpha of 5%, 50 patients are needed (25 per group).

Statistical analysis: Continuous variables will be expressed as means with standard deviations or medians with interquartile ranges (whichever is more appropriate), and discrete variables will be expressed as numbers with percentages. The main efficacy population will consist of all patients being randomized and analyzed according to their original treatment allocation, irrespective of actual received treatment or follow-up (intention-to-treat). The primary comparison will be the mean difference in PImax at month 4. An ANCOVA model will be used to analyze the differences between groups adjusting for baseline PImax. Missing data in the outcomes at month 4 will be imputed by the baseline-observation-carried-forward (BOCF) approach. This will be a conservative method because expected is that patients' PImax will improve after training. For the longitudinal data, a mixed model will be used for repeated measurements including a term for visit, treatment, their interaction, and baseline PImax to account for the correlation within subjects. Similar models will be used for the secondary endpoints. The incidence of adverse events will be summarized by treatment group and in all treatment groups combined in frequency tables, coded according to the introductory guide Medical Dictionary for Regulatory Activities (MedDRA) version 21.0.

Data management: The following measures will be taken to assure the confidentiality and anonymity of the participants' data or documents collected in Castor: a) each participant will be identified in an electronic database by a unique six digit code; b) the list of participant names corresponding to the codes will be stored in a separate encrypted electronic database, safeguarded by the principal investigator; c) only study investigators will have access to the databases and examine individual data or documents; d) all logins will be recorded; e) adopt strict precautions to prevent access to the data or documents by non-authorized persons; f) the handling of data and documents will comply with the General data protection regulation (GDPR) and is further described in the Data Monitoring Plan.

Ethics, dissemination, and safety monitoring: The investigator obtains written informed consent before study participation from participants and from parents if the participant is <16 years old.

The trial is monitored by an external independent party (Julius Clinical). Because of the negligible risk classification minimal monitoring will be necessary. All participants are insured by the sponsor in case of harm due to study participation.

The study will be conducted according to the principles of the Declaration of Helsinki, adapted 19-10-2013, and in accordance with the Medical Research Involving Human Subjects Act (WMO). The code of Conduct as agreed upon 2001 by the Dutch organization of Pediatrics will be used. The study is partly done by minors, which means that in any case of resistance the test and research protocol will be terminated. Resistance means that the patient's behavior obviously differs from or is more excessive compared to participant's normal behavior. The national rules of the Dutch Association of Pediatrics for protection of minor study participants, are followed during the entire study. The results of this study will be publicly disclosed in several publications in peer reviewed scientific journals related to the topic of this study and orally in conferences concerning this theme.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 8 years;
* Respiratory muscle weakness (PImax ≤80 cmH2O (31));
* Maintenance dose (≥2 months) Spinraza® or (≥2 months) Risdiplam or no treatment;
* Given oral and written informed consent when ≥18 years old and additional informed consent by the parents or legal representative if the participant is <16 years old.

Exclusion Criteria:

* Inability to perform respiratory and/or lung-function testing;
* Inability to understand Dutch or English;
* A history of pneumothorax or symptomatic low cardiac output syndrome;
* Treatment period < 2 months of Spinraza® or Risdiplam

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory mouth pressure (PImax) | Baseline
  Maximal inspiratory mouth pressure in Centimeter of Water Column (cmH2O) assessed conform the European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations. Reference values of Wilson et al. 1984 will be used to calculate % of predicted.
Maximal inspiratory mouth pressure (PImax) | 4 months
  Maximal inspiratory mouth pressure in Centimeter of Water Column (cmH2O) assessed conform the European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations. Reference values of Wilson et al. 1984 will be used to calculate % of predicted.
Maximal inspiratory mouth pressure (PImax) | 8 months
  Maximal inspiratory mouth pressure in Centimeter of Water Column (cmH2O) assessed conform the European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations. Reference values of Wilson et al. 1984 will be used to calculate % of predicted.
Maximal inspiratory mouth pressure (PImax) | 12 months
  Maximal inspiratory mouth pressure in Centimeter of Water Column (cmH2O) assessed conform the European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations. Reference values of Wilson et al. 1984 will be used to calculate % of predicted.
Feasibility: adherence from baseline (M0) to 4 months visit (M4) | From baseline (M0) to 4 months visit (M4)
  The completion rate of the estimated number of training sessions over 4 months (>80% of the participants have fulfilled the prescribed treatment = good adherence). Adherence will be monitored by a patient diary, the data saved in the POWERbreathe KHP2 and, two weekly telephone- or video calls by a physiotherapist.
Feasibility: adherence from 4 months (M4) to 8 months visit (M8) | From 4 months (M4) to 8 months visit (M8)
  The completion rate of the estimated number of training sessions over 4 months (>80% of the participants have fulfilled the prescribed treatment = good adherence). Adherence will be monitored by a patient diary, the data saved in the POWERbreathe KHP2 and, two weekly telephone- or video calls by a physiotherapist.
Feasibility: adherence from 8 months (M8) to 12 months visit (M12) | From 8 months (M8) to 12 months visit (M12)
  The completion rate of the estimated number of training sessions over 4 months (>80% of the participants have fulfilled the prescribed treatment = good adherence). Adherence will be monitored by a patient diary, the data saved in the POWERbreathe KHP2 and, two weekly telephone- or video calls by a physiotherapist.
Feasibility: acceptability | 4 months
  The willingness to continue the training (>5 = good acceptability) assessed with a Borg Scale (0-10)
Feasibility: acceptability | 8 months
  The willingness to continue the training (>5 = good acceptability) assessed with a Borg Scale (0-10)
Feasibility: acceptability | 12 months
  The willingness to continue the training (>5 = good acceptability) assessed with a Borg Scale (0-10)

SECONDARY OUTCOMES:
Maximal expiratory mouth pressure (PEmax) | Baseline
  Maximal expiratory mouth pressure in Centimeter of Water Column (cmH2O) assessed conform the European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations. Reference values of Wilson et al. 1984 will be used to calculate % of predicted.
Maximal expiratory mouth pressure (PEmax) | 4 months
  Maximal expiratory mouth pressure in Centimeter of Water Column (cmH2O) assessed conform the European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations. Reference values of Wilson et al. 1984 will be used to calculate % of predicted.
Maximal expiratory mouth pressure (PEmax) | 8 months
  Maximal expiratory mouth pressure in Centimeter of Water Column (cmH2O) assessed conform the European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations. Reference values of Wilson et al. 1984 will be used to calculate % of predicted.
Maximal expiratory mouth pressure (PEmax) | 12 months
  Maximal expiratory mouth pressure in Centimeter of Water Column (cmH2O) assessed conform the European Respiratory Society/American Thoracic Society (ERS/ATS) recommendations. Reference values of Wilson et al. 1984 will be used to calculate % of predicted.
Health related quality of life | Baseline
  Health related quality of life will be measured with the 36-item Short Form Health Survey (SF36) for adults and the Pediatric Quality of Life Inventory (PedsQL) for children and their parents/caregivers.
Health related quality of life | 4 months
  Health related quality of life will be measured with the 36-item Short Form Health Survey (SF36) for adults and the Pediatric Quality of Life Inventory (PedsQL) for children and their parents/caregivers.
Health related quality of life | 8 months
  Health related quality of life will be measured with the 36-item Short Form Health Survey (SF36) for adults and the Pediatric Quality of Life Inventory (PedsQL) for children and their parents/caregivers.
Health related quality of life | 12 months
  Health related quality of life will be measured with the 36-item Short Form Health Survey (SF36) for adults and the Pediatric Quality of Life Inventory (PedsQL) for children and their parents/caregivers.
Forced vital capacity (FVC) | Baseline
  Forced vital capacity in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Forced vital capacity (FVC) | 4 months
  Forced vital capacity in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Forced vital capacity (FVC) | 8 months
  Forced vital capacity in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Forced vital capacity (FVC) | 12 months
  Forced vital capacity in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Slow vital capacity (SVC) | Baseline
  Slow vital capacity in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Slow vital capacity (SVC) | 4 months
  Slow vital capacity in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Slow vital capacity (SVC) | 8 months
  Slow vital capacity in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Slow vital capacity (SVC) | 12 months
  Slow vital capacity in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Peak expiratory flow (PEF) | Baseline
  Peak expiratory flow in liters per second assessed conform the ERS/ATS recommendations. Reference values of Quanjer et al. 1993 will be used to calculate % of predicted for adults and Koopman et al. 2011 will be used to calculate % of predicted for kids.
Peak expiratory flow (PEF) | 4 months
  Peak expiratory flow in liters per second assessed conform the ERS/ATS recommendations. Reference values of Quanjer et al. 1993 will be used to calculate % of predicted for adults and Koopman et al. 2011 will be used to calculate % of predicted for kids.
Peak expiratory flow (PEF) | 8 months
  Peak expiratory flow in liters per second assessed conform the ERS/ATS recommendations. Reference values of Quanjer et al. 1993 will be used to calculate % of predicted for adults and Koopman et al. 2011 will be used to calculate % of predicted for kids.
Peak expiratory flow (PEF) | 12 months
  Peak expiratory flow in liters per second assessed conform the ERS/ATS recommendations. Reference values of Quanjer et al. 1993 will be used to calculate % of predicted for adults and Koopman et al. 2011 will be used to calculate % of predicted for kids.
Forced expiratory volume in 1 second (FEV1) | Baseline
  Forced expiratory volume in 1 second in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Forced expiratory volume in 1 second (FEV1) | 4 months
  Forced expiratory volume in 1 second in liters assessed conform the ERS/ATS recommendations.Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Forced expiratory volume in 1 second (FEV1) | 8 months
  Forced expiratory volume in 1 second in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Forced expiratory volume in 1 second (FEV1) | 12 months
  Forced expiratory volume in 1 second in liters assessed conform the ERS/ATS recommendations. Reference values from Quanjer et al. 2012 will be used to calculate % of predicted.
Peak cough flow (PCF) | Baseline
  Peak cough flow in liters per second assessed conform the ERS/ATS recommendations.
Peak cough flow (PCF) | 4 months
  Peak cough flow in liters per second assessed conform the ERS/ATS recommendations.
Peak cough flow (PCF) | 8 months
  Peak cough flow in liters per second assessed conform the ERS/ATS recommendations.
Peak cough flow (PCF) | 12 months
  Peak cough flow in liters per second assessed conform the ERS/ATS recommendations.
Sniff Nasal Inspiratory Pressure (SNIP) | Baseline
  Sniff Nasal Inspiratory Pressure in Kilopascal (kPa) assessed conform the ERS/ATS recommendations.
Sniff Nasal Inspiratory Pressure (SNIP) | 4 months
  Sniff Nasal Inspiratory Pressure in Kilopascal (kPa) assessed conform the ERS/ATS recommendations.
Sniff Nasal Inspiratory Pressure (SNIP) | 8 months
  Sniff Nasal Inspiratory Pressure in Kilopascal (kPa) assessed conform the ERS/ATS recommendations.
Sniff Nasal Inspiratory Pressure (SNIP) | 12 months
  Sniff Nasal Inspiratory Pressure in Kilopascal (kPa) assessed conform the ERS/ATS recommendations.
Mouth occlusion pressure at 100ms (P0.1) | Baseline
  Mouth occlusion pressure at 100ms during quiet breathing in Kilopascal (kPa). P0.1 is a marker of neuromuscular ventilator drive, which is independent of the patient's effort. Assessed conform the ERS/ATS recommendations. Reference values of Criee 2003 will be used to calculate % of predicted.
Mouth occlusion pressure at 100ms (P0.1) | 4 months
  Mouth occlusion pressure at 100ms during quiet breathing in Kilopascal (kPa). P0.1 is a marker of neuromuscular ventilator drive, which is independent of the patient's effort. Assessed conform the ERS/ATS recommendations. Reference values of Criee 2003 will be used to calculate % of predicted.
Mouth occlusion pressure at 100ms (P0.1) | 8 months
  Mouth occlusion pressure at 100ms during quiet breathing in Kilopascal (kPa). P0.1 is a marker of neuromuscular ventilator drive, which is independent of the patient's effort. Assessed conform the ERS/ATS recommendations. Reference values of Criee 2003 will be used to calculate % of predicted.
Mouth occlusion pressure at 100ms (P0.1) | 12 months
  Mouth occlusion pressure at 100ms during quiet breathing in Kilopascal (kPa). P0.1 is a marker of neuromuscular ventilator drive, which is independent of the patient's effort. Assessed conform the ERS/ATS recommendations. Reference values of Criee 2003 will be used to calculate % of predicted.
P0.1/PImax | Baseline
  The ratio of P0.1/PImax have been suggested as important predictor of impending respiratory muscle fatigue (work of breathing)
P0.1/PImax | 4 months
  The ratio of P0.1/PImax have been suggested as important predictor of impending respiratory muscle fatigue (work of breathing)
P0.1/PImax | 8 months
  The ratio of P0.1/PImax have been suggested as important predictor of impending respiratory muscle fatigue (work of breathing)
P0.1/PImax | 12 months
  The ratio of P0.1/PImax have been suggested as important predictor of impending respiratory muscle fatigue (work of breathing)
Medical Research Council (MRC) dyspnea scale | Baseline
  This scale measures perceived respiratory disability.
Medical Research Council (MRC) dyspnea scale | 4 months
  This scale measures perceived respiratory disability.
Medical Research Council (MRC) dyspnea scale | 8 months
  This scale measures perceived respiratory disability.
Medical Research Council (MRC) dyspnea scale | 12 months
  This scale measures perceived respiratory disability.
Respiratory infections | Assessed during the two weekly telephone consultations.
  Respiratory infection frequency (based on the need for antibiotics and/or hospitalization).
Respiratory infections | Assessed during the 4 months visit.
  Respiratory infection frequency (based on the need for antibiotics and/or hospitalization).
Respiratory infections | Assessed during the 8 months visit.
  Respiratory infection frequency (based on the need for antibiotics and/or hospitalization).
Respiratory infections | Assessed during the 12 months visit.
  Respiratory infection frequency (based on the need for antibiotics and/or hospitalization).
Adverse Events | During the whole 12 months.
  Adverse Events
  Adverse Events
  Adverse Events Adverse Events coded according to the introductory guide MedDRA version 21.0
Dyspnea immediately after lung function measure and after each training session | After each training session
  Assesses with a Borg scale ranging from 0-10.
Dyspnea immediately after lung function measure and after each training session | Baseline
  Assesses with a Borg scale ranging from 0-10.
Dyspnea immediately after lung function measure and after each training session | 4 months
  Assesses with a Borg scale ranging from 0-10.
Dyspnea immediately after lung function measure and after each training session | 8 months
  Assesses with a Borg scale ranging from 0-10.
Dyspnea immediately after lung function measure and after each training session | 12 months
  Assesses with a Borg scale ranging from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hulzebos, Dr, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wadman RI, Vrancken AF, van den Berg LH, van der Pol WL. Dysfunction of the neuromuscular junction in spinal muscular atrophy types 2 and 3. Neurology. 2012 Nov 13;79(20):2050-5. doi: 10.1212/WNL.0b013e3182749eca. Epub 2012 Oct 31. PMID 23115209
- [Background] Finkel RS, Sejersen T, Mercuri E; ENMC SMA Workshop Study Group. 218th ENMC International Workshop:: Revisiting the consensus on standards of care in SMA Naarden, The Netherlands, 19-21 February 2016. Neuromuscul Disord. 2017 Jun;27(6):596-605. doi: 10.1016/j.nmd.2017.02.014. Epub 2017 Mar 2. No abstract available. PMID 28392274
- [Background] Lunn MR, Wang CH. Spinal muscular atrophy. Lancet. 2008 Jun 21;371(9630):2120-33. doi: 10.1016/S0140-6736(08)60921-6. PMID 18572081
- [Background] Verhaart IEC, Robertson A, Wilson IJ, Aartsma-Rus A, Cameron S, Jones CC, Cook SF, Lochmuller H. Prevalence, incidence and carrier frequency of 5q-linked spinal muscular atrophy - a literature review. Orphanet J Rare Dis. 2017 Jul 4;12(1):124. doi: 10.1186/s13023-017-0671-8. PMID 28676062
- [Background] Wang CH, Finkel RS, Bertini ES, Schroth M, Simonds A, Wong B, Aloysius A, Morrison L, Main M, Crawford TO, Trela A; Participants of the International Conference on SMA Standard of Care. Consensus statement for standard of care in spinal muscular atrophy. J Child Neurol. 2007 Aug;22(8):1027-49. doi: 10.1177/0883073807305788. PMID 17761659
- [Background] Stam M, Wadman RI, Wijngaarde CA, Bartels B, Asselman FL, Otto LAM, Goedee HS, Habets LE, de Groot JF, Schoenmakers MAGC, Cuppen I, van den Berg LH, van der Pol WL. Protocol for a phase II, monocentre, double-blind, placebo-controlled, cross-over trial to assess efficacy of pyridostigmine in patients with spinal muscular atrophy types 2-4 (SPACE trial). BMJ Open. 2018 Jul 30;8(7):e019932. doi: 10.1136/bmjopen-2017-019932. PMID 30061431
- [Background] Mongiovi P, Dilek N, Garland C, Hunter M, Kissel JT, Luebbe E, McDermott MP, Johnson N, Heatwole C. Patient Reported Impact of Symptoms in Spinal Muscular Atrophy (PRISM-SMA). Neurology. 2018 Sep 25;91(13):e1206-e1214. doi: 10.1212/WNL.0000000000006241. Epub 2018 Aug 24. PMID 30143566
- [Background] Bartels B, Habets LE, Stam M, Wadman RI, Wijngaarde CA, Schoenmakers MAGC, Takken T, Hulzebos EHJ, van der Pol WL, de Groot JF. Assessment of fatigability in patients with spinal muscular atrophy: development and content validity of a set of endurance tests. BMC Neurol. 2019 Feb 9;19(1):21. doi: 10.1186/s12883-019-1244-3. PMID 30738436
- [Background] Bartels B, de Groot JF, Habets LE, Wijngaarde CA, Vink W, Stam M, Asselman FL, van Eijk RPA, van der Pol WL. Fatigability in spinal muscular atrophy: validity and reliability of endurance shuttle tests. Orphanet J Rare Dis. 2020 Mar 23;15(1):75. doi: 10.1186/s13023-020-1348-2. PMID 32293503
- [Background] Wadman RI, Wijngaarde CA, Stam M, Bartels B, Otto LAM, Lemmink HH, Schoenmakers MAGC, Cuppen I, van den Berg LH, van der Pol WL. Muscle strength and motor function throughout life in a cross-sectional cohort of 180 patients with spinal muscular atrophy types 1c-4. Eur J Neurol. 2018 Mar;25(3):512-518. doi: 10.1111/ene.13534. Epub 2018 Feb 2. PMID 29194869
- [Background] Finkel RS, Mercuri E, Darras BT, Connolly AM, Kuntz NL, Kirschner J, Chiriboga CA, Saito K, Servais L, Tizzano E, Topaloglu H, Tulinius M, Montes J, Glanzman AM, Bishop K, Zhong ZJ, Gheuens S, Bennett CF, Schneider E, Farwell W, De Vivo DC; ENDEAR Study Group. Nusinersen versus Sham Control in Infantile-Onset Spinal Muscular Atrophy. N Engl J Med. 2017 Nov 2;377(18):1723-1732. doi: 10.1056/NEJMoa1702752. PMID 29091570
- [Background] Paul GR, Gushue C, Kotha K, Shell R. The respiratory impact of novel therapies for spinal muscular atrophy. Pediatr Pulmonol. 2021 Apr;56(4):721-728. doi: 10.1002/ppul.25135. Epub 2020 Nov 2. PMID 33098622
- [Background] Heitschmidt L, Pichlmaier L, Eckerland M, Steindor M, Olivier M, Fuge I, Kolbel H, Hirtz R, Stehling F. Nusinersen does not improve lung function in a cohort of children with spinal muscular atrophy - A single-center retrospective study. Eur J Paediatr Neurol. 2021 Mar;31:88-91. doi: 10.1016/j.ejpn.2021.02.007. Epub 2021 Feb 28. PMID 33711791
- [Background] Koessler W, Wanke T, Winkler G, Nader A, Toifl K, Kurz H, Zwick H. 2 Years' experience with inspiratory muscle training in patients with neuromuscular disorders. Chest. 2001 Sep;120(3):765-9. doi: 10.1378/chest.120.3.765. PMID 11555507
- [Background] Winkler G, Zifko U, Nader A, Frank W, Zwick H, Toifl K, Wanke T. Dose-dependent effects of inspiratory muscle training in neuromuscular disorders. Muscle Nerve. 2000 Aug;23(8):1257-60. doi: 10.1002/1097-4598(200008)23:83.0.co;2-m. PMID 10918264
- [Background] Aslan GK, Gurses HN, Issever H, Kiyan E. Effects of respiratory muscle training on pulmonary functions in patients with slowly progressive neuromuscular disease: a randomized controlled trial. Clin Rehabil. 2014 Jun;28(6):573-81. doi: 10.1177/0269215513512215. Epub 2013 Nov 25. PMID 24275453
- [Background] Human A, Morrow BM. Inspiratory muscle training in children and adolescents living with neuromuscular diseases: A pre-experimental study. S Afr J Physiother. 2021 Aug 31;77(1):1577. doi: 10.4102/sajp.v77i1.1577. eCollection 2021. PMID 34522820
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Background] Koopman M, Zanen P, Kruitwagen CL, van der Ent CK, Arets HG. Reference values for paediatric pulmonary function testing: The Utrecht dataset. Respir Med. 2011 Jan;105(1):15-23. doi: 10.1016/j.rmed.2010.07.020. PMID 20889322
- [Background] Criee CP; German Airway League. [Recommendations of the German Airway League (Deutsche Atemwegsliga) for the determination of inspiratory muscle function]. Pneumologie. 2003 Feb;57(2):98-100. doi: 10.1055/s-2003-37154. No abstract available. German. PMID 12579465
- [Background] Wilson SH, Cooke NT, Edwards RH, Spiro SG. Predicted normal values for maximal respiratory pressures in caucasian adults and children. Thorax. 1984 Jul;39(7):535-8. doi: 10.1136/thx.39.7.535. PMID 6463933
- [Derived] Kant-Smits K, Bartels B, Asselman FL, Veldhoen ES, van Eijk RPA, van der Pol WL, Hulzebos EHJ. The RESISTANT study (Respiratory Muscle Training in Patients with Spinal Muscular Atrophy): study protocol for a randomized controlled trial. BMC Neurol. 2023 Mar 23;23(1):118. doi: 10.1186/s12883-023-03136-3. PMID 36959618